CLINICAL TRIAL: NCT02941133
Title: Effectiveness of Neural Mobilization Techniques Compared to Standard Care Treatment in Patients With Lumbar Radiculitis: A Randomized Clinical Trial
Brief Title: Comparison of Neural Mobilization Techniques to Standard Care Treatment in Patients With Lumbar Radiculitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Michalis Efstathiou (Other)
Responsible Party: Sponsor-Investigator, Michalis Efstathiou, Assosiate Lecturer, University of Nicosia
Organization: University of Nicosia (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MISS13
Record Dates: First submitted 2016-10-19; First posted 2016-10-21 (Estimated); Last update posted 2017-05-05 (Actual); Status verified 2017-05

CONDITIONS: Radiculitis
MeSH Terms: conditions — Radiculopathy | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neural Mobilization Group (Experimental): Patients in this group will be treated with neural mobilization techniques.
  Interventions: Other: Neural Mobilization
- Standard Care Group (Experimental): Patients in this group will be treated with standard care (ultrasound, exercise, TENS, massage)
  Interventions: Other: Standard Care

INTERVENTIONS:
Other: Neural Mobilization — Neural mobilization techniques aimed at the lumbar root that is affected
  Arms: Neural Mobilization Group
Other: Standard Care — Ultrasound - Transcutaneous electrical nerve stimulation (TENS) - Massage therapy - Strengthening exercises
  Arms: Standard Care Group

SUMMARY:
The purpose of this study is to determine the effectiveness of neural mobilization techniques compared to standard care treatment in patients with lumbar radiculitis.

DETAILED DESCRIPTION:
Background:

Radicular pain has been regarded as a distinct pain entity as its pathophysiology differs from that of somatic referred pain and nociceptive pain. Radicular lumbar pain describes sensitized nerve roots of the lumbar spine or peripheral nerve trunks that are capable of producing pain (usually below the knee) and/or other symptoms in the absence of true nerve tissue damage. This type of pain is evoked by ectopic discharges stemming from lumbar dorsal roots or their ganglions. The most common causes for this type of pain is the inflammatory environment that is produced by substances contained in the herniated material of injured lumbar intervertebral discs.

It has been suggested that patients presenting with functional (e.g. mechanosensitivity) but not structural nerve root problems, can be identified through screening and further classified as a discrete group of patients that benefit from specific neural mobilization techniques.

Neural mobilization techniques have gained considerable amount of attention amongst therapists and researchers for the assessment and treatment of painful conditions that occasionally involve a neural element in their pathophysiology such as lumbar radicular pain. Studies exploring the effect of neural mobilization techniques on patients with lumbar radicular pain have generally shown good results but they are lacking in adequate sample size and methodological quality.

The aim of this study is to compare the effectiveness of neural mobilization techniques to standard care physiotherapy treatment (ultrasound, general exercises, massage therapy, transcutaneous electrical nerve stimulation) in patients with lumbar radiculitis.

Participants:

Patients with low back pain that radiates to the lower limb.

Patients that satisfy the inclusion criteria will be screened and classified by another researcher into the distinct group of lumbar radiculitis. Another researcher will take baseline measurements and all patients of this sub-group will be randomly assigned to receive either neural mobilization or standard care physiotherapy treatment. Both groups will receive a total of 10 treatments twice per week for 5 weeks. Patients will be assessed using specific outcome measures prior to treatment (baseline), at 5 weeks (post treatment) and 6 months after treatment.

Statistical analysis:

Data will be analysed with the Statistical Package for the Social Sciences (SPSS), version 22. Intension to treat analysis will be applied. A two-way mixed-model analysis of variance will be used for outcome measures, with treatment groups (neural mobilization or standard care treatment) as the between-subject variable and time (baseline, 1 month follow up, six months follow up) as the within-subject variable. Comparison of baseline demographic characteristics will be analysed using the t-tests for continuous variables and the chi square tests for categorical variables.

ELIGIBILITY:
Inclusion Criteria:

* Patients with low back pain and pain that radiates in the lower limb
* Duration of symptoms > 6 weeks
* Patients willing to be reassessed after 6 months
* Patients willing to give written informed consent

Exclusion Criteria:

* History of spinal surgery
* History of surgery or injury in the lower limbs in the past 6 months
* Signs and symptoms of central nervous system involvement
* Nerve root blocks for the past 6 weeks
* History of diabetes
* History of polyneuropathies
* History of vascular pathologies in the lower limbs
* History of systemic pathologies
* History of inflammatory arthropathies

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2017-09 (Estimated); Primary Completion 2020-03 (Estimated); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale (VAS) - Measure assessing change | Change from baseline after 5 weeks and at 6 months
  The VAS is a 100-point pain assessment scale ranging from 0 (no pain) to 100 (worst pain possible).

SECONDARY OUTCOMES:
Roland Morris Disability Questionnaire (RMDQ) - Measure assessing change | Change from baseline after 5 weeks and at 6 months
  The questioner measures the level of patients' disability.
Fear Avoidance and Beliefs Questionnaire (FABQ) - Measure assessing change | Change from baseline after 5 weeks and at 6 months
  The questioner evaluates fear-avoidance beliefs of patients with low back pain in the clinical setting.
Handheld dynamometer - Measure assessing change | Change from baseline after 5 weeks and at 6 months
  Changes in Muscle Strength assessed with the handheld dynamometer

CONTACTS AND LOCATIONS:
Overall Officials: Michalis Efstathiou, MSc, Principal Investigator — University of Nicosia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Schafer A, Hall T, Muller G, Briffa K. Outcomes differ between subgroups of patients with low back and leg pain following neural manual therapy: a prospective cohort study. Eur Spine J. 2011 Mar;20(3):482-90. doi: 10.1007/s00586-010-1632-2. Epub 2010 Dec 1. PMID 21116662